CLINICAL TRIAL: NCT02399137
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study of MM-141 Plus Nab-paclitaxel and Gemcitabine Versus Nab-paclitaxel and Gemcitabine in Front-line Metastatic Pancreatic Cancer
Brief Title: A Phase 2 Study of MM-141 Plus Nab-paclitaxel and Gemcitabine in Front-line Metastatic Pancreatic Cancer
Acronym: CARRIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MM-141-07-02-02
Record Dates: First submitted 2015-03-19; First posted 2015-03-26 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Front-line Pancreatic Cancer; Metastatic Pancreatic Cancer; Gemcitabine; Nab-paclitaxel; Abraxane; Free IGF-1; Heregulin
MeSH Terms: conditions — Pancreatic Neoplasms; Fibromatosis, Gingival, 2 | interventions — Istiratumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental Arm) (Experimental): MM-141 in combination with nab-paclitaxel and gemcitabine
  Interventions: Drug: MM-141; Drug: Gemcitabine; Drug: Nab-Paclitaxel
- Arm B (Comparator Arm) (Active Comparator): Placebo in combination with nab-paclitaxel and gemcitabine
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Nab-Paclitaxel
- Observational Group (No Intervention)

INTERVENTIONS:
Drug: MM-141
  Arms: Arm A (Experimental Arm)
Drug: Placebo
  Arms: Arm B (Comparator Arm)
Drug: Gemcitabine
  Other Names: Gemzar
  Arms: Arm A (Experimental Arm); Arm B (Comparator Arm)
Drug: Nab-Paclitaxel
  Other Names: Abraxane
  Arms: Arm A (Experimental Arm); Arm B (Comparator Arm)

SUMMARY:
The purpose of this study is to determine whether the combination of MM-141 plus nab-paclitaxel and gemcitabine is more effective than nab-paclitaxel and gemcitabine alone based on Progression Free Survival (PFS) in front-line metastatic pancreatic cancer patients with high serum levels of free IGF-1.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 2 study of MM-141 plus nab-paclitaxel and gemcitabine or placebo plus nab-paclitaxel and gemcitabine in front-line metastatic pancreatic cancer. All patients will be initially screened for free IGF-1 status. Eligible patients with high free IGF-1 will be randomized to receive MM-141 plus nab-paclitaxel and gemcitabine or placebo plus nab-paclitaxel and gemcitabine and patients. Patients with low free IGF-1 or patients who have high free IGF-1 but are not otherwise eligible will be followed in an observational group.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic adenocarcinoma of the pancreas. Patients with islet cell neoplasms are not eligible.
* Patient must have received no prior radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of metastatic disease.
* Blood sample sent for free IGF-1 testing
* ECOG performance status (PS) of 0 or 1

Exclusion Criteria:

* Patients who only present with localized disease
* Patients with CNS malignancies (primary or metastatic)
* Clinically significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-05; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Approximately 2 years

SECONDARY OUTCOMES:
Overall Survival | Approximately 2.5 years
Objective Response Rate according to RECIST v1.1 | Approximately 2 years
Duration of Response according to RECIST v1.1 | Approximately 2 years
Rate of adverse events reported with the combination of MM-141 with nab-paclitaxel and gemcitabine versus the comparator arm | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MM-141 Medical Director, MD, Study Director — Merrimack Pharmaceuticals
Locations (66):
- United States (47):
  - Banner MD Anderson Cancer Ctr., Gilbert, Arizona
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - UCLA School of Medicine, Los Angeles, California
  - Cancer Care Assoc Med Grp, Redondo Beach, California
  - UCSF Cancer Center, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Central Coast Med Onc Corp, Santa Maria, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Baptist Health Med Gr Onc, LLC, Miami, Florida
  - Florida Cancer AffiliatesOcala, Ocala, Florida
  - Memorial Regional Hospital, Pembroke Pines, Florida
  - Cancer Treatment Centers of America-Georgia, Newnan, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Illinois Cancer Specialists, Chicago, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Midwest Regional Medical Cntr, Zion, Illinois
  - Nylen Cancer Center, Sioux City, Iowa
  - Cancer Center of Acadiana Research Department, Lafayette, Louisiana
  - Reliant Medical Group, Inc., Worcester, Massachusetts
  - Compr Cancer Centers of Nevada, Henderson, Nevada
  - New York Oncology HematologyPC, Albany, New York
  - Roswell Park Cancer Inst, Buffalo, New York
  - Bassett Cancer Institute, Cooperstown, New York
  - North Shore Hematology Oncology Associates, PC, East Setauket, New York
  - Columbia University Medical Center, New York, New York
  - Columbia University, New York, New York
  - Mid Ohio Onco/ Zangmeister Ctr, Columbus, Ohio
  - Tulsa Cancer Institute, PLLC, Tulsa, Oklahoma
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology P A Bedford, Bedford, Texas
  - Texas Oncology-Dallas P.H., Dallas, Texas
  - Brooke Army Medical Center (BAMC), Fort Sam Houston, Texas
  - Texas Oncology-Paris, Paris, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Texas Oncology SA Medical Ctr, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Virginia Cancer Specialists PC, Fairfax, Virginia
  - Onc and Hem Asso of SW VA Inc, Salem, Virginia
  - Cancer Care Northwest, P.S., Spokane Valley, Washington
  - Northwest Cancer SpecialistsPC, Vancouver, Washington
- Cross Cancer Institute, Edmonton, Alberta, Canada
- Germany (5):
  - Klinikum rechts der Isar - TUM, München, Bavaria
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Caritasklinik St. Theresia, Saarbrücken, Saarland
  - Vivantes Klinikum Neukoelln, Berlin
  - Charite Universitaetsmd Berlin, Berlin
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - WSZ im. L. Rydygiera wToruniu, Torun
- Spain (6):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital U de Fuenlabrada, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (5):
  - Guy's Hospital, London, Greater London
  - Sarah Cannon Research Institute UK, London, Greater London
  - The Christie, Manchester, Greater Manchester
  - Royal Marsden Hospital, Sutton, Surrey
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Kundranda M, Gracian AC, Zafar SF, Meiri E, Bendell J, Algul H, Rivera F, Ahn ER, Watkins D, Pelzer U, Charu V, Zalutskaya A, Kuesters G, Pipas JM, Santillana S, Askoxylakis V, Ko AH. Randomized, double-blind, placebo-controlled phase II study of istiratumab (MM-141) plus nab-paclitaxel and gemcitabine versus nab-paclitaxel and gemcitabine in front-line metastatic pancreatic cancer (CARRIE). Ann Oncol. 2020 Jan;31(1):79-87. doi: 10.1016/j.annonc.2019.09.004. PMID 31912800